CLINICAL TRIAL: NCT04914130
Title: A Prospective, Observational Study to Examine the Effects of Ageing on the Clinical Outcomes of People Living With HIV in South Korea
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0853
Record Dates: First submitted 2021-05-24; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: HIV Infection
Keywords: HIV; Aging; Comorbidity; non-communicable diseases
MeSH Terms: conditions — HIV Infections; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood (up to 91ml for the HIV positive group and 73ml in the HIV negative group)
  * Urine sample (20 - 30 mL)
  * Stool sample (2 or 3 scoops)
  * Plus storage samples collected during the lumbar puncture, as described in section 8.5 All samples for storage will be collected at the clinic; however the stool sample may be collected by the subject at home. In this case the subject will be provided with a container without medium and advised to collect two to three scoops of faeces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Older HIV-positive cohort (n=500): * documented HIV infection
  * age >50 years at study entry
  * Korean ethnicity
  * likely route of HIV acquisition via sexual exposure by male to male exposure
  * able to comprehend study patient information leaflet.
  * Virologically suppressed subjects Subjects with primary HIV infection are eligible and investigators are encouraged to recruit such subjects. Our target population (those infected with HIV via sexual routes of men who have sex with men) has been chosen as this group represent the vast majority of older HIV-positive individuals attending for care in Korea; analyses of other groups (e.g. injection drug users, those infected through blood/blood products and transgender individuals), who may have very different needs and outcomes, would likely be under-powered.
  Interventions: Other: Study specific testing procedures
- Younger HIV-positive cohort (n=250): * documented HIV infection
  * age <50 at study entry*
  * Korean ethnicity
  * likely route of HIV acquisition via sexual exposure by male to male exposure
  * able to comprehend study patient information leaflet * this group will comprise of at least 70 subjects in each of the following age groups: 20-29, 30-39, 40-49 years. Recruitment will be monitored by the Study Monitoring Team
  Interventions: Other: Study specific testing procedures
- HIV-negative cohort (n=250): * documented negative HIV test at screening
  * age >50 years at study entry
  * Korean ethnicity
  * self reported sexual preferences of men who have sex with men
  To enroll matched control, we will try to match age, sexual orientation, and participating clinic.
  Interventions: Other: Study specific testing procedures

INTERVENTIONS:
Other: Study specific testing procedures — Study specific procedures includes blood sampling, neurocognitive testing, respiratory questionnaire, brain MRI for MRI substudy group, lumbar puncture for MRI substudy group, etc

SUMMARY:
This study is to investigate how HIV affects ageing process, especially in Asian populations in various organ system, including brain, kidney, liver and etc. There are some articles that describing the ageing process in PWHIV, but there has been a limited number of articles that comparing ageing process by ethnicities. And the endpoints of those limited number of articles are including more general variables like all-cause mortality, detectable viral load and days to regimen changes. There is no extensive study of ageing by function of each organ system in Asia. This proposal contains more specific observation points on function/dysfxn of each organ system, especially for brain function as an MRI sub-study. The MRI sub-study has a large portion of this proposal as analysis of the neurocognitive function in HIV ageing, which has not been extensively studied in Asia, nor it hasn't been compared to other ethnic groups.

With this proposal, we can see if there are differences by ethnicities compared to POPPY/COBRA results, and even if there are no differences, we can increase the number and diversify of cohort subjects and strengthen the level of evidence of cohort study.

Our study, by enrolling both younger and older HIV-positive individuals with a matched HIV-negative control group, will be in the unique position to determine the effects of ageing and HIV status on chronic HIV-infection. In addition, results from this study will be well placed to assist in informing future HIV treatment guidelines on the monitoring of chronic HIV infection in older subjects and assisting in the design of future interventional studies for the treatment of age associated co-morbidities.

DETAILED DESCRIPTION:
Study Design: Multicentre, prospective, observational study over 3 years. Our study will describe the impact of advancing age on the experience of living with HIV in South Korea. To address this we will establish cohorts of HIV-positive people aged >50 and <50 years as well as demographically matched HIV-negative people aged >50 years. Although 2 years of follow up duration is short period to evaluate the effect of aging, this period could give us an insights for necessity of longer follow up study.

Setting:

Subjects will be recruited from three clinics: Severance Hospital; Seoul Medical Center; National Medical Center.

Number of Patients: Older HIV-positive cohort (n=500); Younger HIV-positive cohort (n=250); HIV-negative cohort (n=250). We arbitrarily decided these numbers of subjects considering the numbers of subjects of POPPY-UK study (1000, 500, and 500 subjects, respectively), feasibility of recruitment, and possible budget. Our choice of sample size is largely pragmatic, reflecting the number of older patients receiving care and the proportion that are expected to participate. Detailed sample size calculations are difficult given the wide range of topics and methodological approaches proposed.

Sample size was chosen pragmatically based on

1) the number of HIV pts of three participating hospitals (NMC≒1200, severance≒700, SMC≒300) 2) feasibility of recruitment 3) and possible budget

1. Screening

   Each subject must sign an Informed Consent Form prior to the conduct of any screening procedures.

   The purpose of the screening visit is to evaluate that the subject meets study inclusion/exclusion criteria. HIV antibody testing will be undertaken for subjects undergoing screening for the HIV-negative cohort.
2. Visit 1 (Baseline visit)

   The baseline visit will perform evaluations as per schedule of visits.

   The baseline visit is expected to take 1-2 hours; if possible the subject should attend fasted. The following information will be collected:

   • Baseline demographics: age; sex; sexual orientation; date of birth; education.

   • Socio-economic status: employment; household dependents; household income; housing.

   • Quality of life questionnaire.

   • Anthropometrics: height; weight; body mass index; waist circumference.

   • Lifestyle factors: current/past cigarette smoking; alcohol use; recreational drug use.

   • Full clinical history: to include cardiovascular events (hypertension, myocardial infarction, angina or acute coronary syndromes, cardiogenic arrhythmias, coronary artery stenting/bypass grafting, peripheral vascular disease), renal failure, liver failure, diabetes, malignancies, falls, fractures, joint disease or joint replacements.

   • Simple measurement of walking speed over a distance of 15 feet (457 cms).

   • Blood pressure will be estimated using an automated device.

   • Family medical history: to include any cardiovascular disease, type 2 diabetes mellitus, malignancies, mental illness, dementia or Alzheimer's disease, parental hip fractures.

   • Current and recent (over past 12 months) antiretroviral use: type of antiretroviral; start/stop dates; dose; frequency of dosing; side effects; reasons for prior changes/discontinuations.

   • Duration of HIV infection and date of HIV-seroconversion if known
   * Adherence assessment
   * Use of any other medications (including, but not limited to, anti-hypertensives, anti-depressants, vitamin D and/or calcium replacement therapy, lipid-lowering drugs, regular use of analgesics, herbal remedies, other over-the-counter drugs): type of drug; start/stop dates; dose; frequency of dosing; side effects.
   * Neurocognitive function: specific memory and cognitive testing assessing cortical and sub-cortical function.
   * Pain assessment: regional and widespread pain collected using a validated mannequin; nature of onset; duration; intensity; resulting disability
   * Falls risk (study questionnaire)
   * Fracture risk (study questionnaire)
   * Frailty assessment (study questionnaire)
   * Most recent laboratory tests will be recorded (assessed in the HIV-negative cohort): renal, liver, lipid and bone profiles, glucose, full blood count, sexual health screen, hepatitis C serology. These tests should have been performed within a year of the clinic visit.
   * Blood (serum, plasma, and PBMC) and urine samples: stored for subsequent projects of the potential pathogenic mechanisms underlying age-related diseases. This will include assessment of vitamin-D and PTH
   * Blood (plasma) will be collected for pharmacokinetic analysis (including but not limited to antiretroviral drug exposure)
3. Visit 2 (1st year follow up visit)

   This follow up visit will be performed as per schedule of visits. Only HIV-positive cohorts will be invited to undertake this visit with this visit expected to take 1 hour.

   The following will be assessed:
   * Changes to lifestyle and socio-economic status over the past year.
   * Significant clinical events occurring over the past year: dates of onset and resolution, use of medical services, changes to antiretroviral and other medications, and resulting ongoing health concerns.
   * Blood pressure will be estimated using an automated device.
   * Details of access to health care services over the past year: visits to hospital, and medical investigations performed (information obtained by direct questioning and through medical records review).
   * Most recent laboratory tests will be recorded: renal, liver, lipid and bone profiles, glucose, full blood count, sexual health screen, hepatitis C serology (Within the past year)
   * Concomitant medications: start/stop dates; dose; dosing frequency; side effects.
   * Fracture occurrence and fracture risk (see study questionnaire in appendix 1)
   * Regional and widespread pain.

3a Visit 2 (1st year follow up visit) for HIV negative participants.

These participants will be contacted by telephone by arrangement with the study nurse. They may be asked to attend the clinic in order to facilitate this visit.

Details of any changes in circumstances or illnesses and medication will be documented.

4 Visit 3 (2nd year follow up visit)

This follow up visit will be performed as per schedule of visits (2.0).

This visit is expected to take 1-2 hours; if possible the subject should attend fasted. The following information will be collected:

* Changes to lifestyle and socio-economic status over the past year.
* Significant clinical events occurring over the past year: dates of onset and resolution, use of medical services, treatments, and resulting ongoing health concerns.
* Details of access to health care services over the past year: visits to hospital, and medical investigations performed (information obtained by direct questioning and through medical records review).
* Simple measurement of walking speed over a distance of 15 feet (457 cms).
* Blood pressure will be estimated using an automated device.
* Concomitant medications: start/stop dates; dose; dosing frequency; side effects.
* Fracture occurrence and fracture risk (see study questionnaire in appendix 1).
* Neurocognitive function: specific memory and cognitive testing assessing cortical and sub-cortical function.
* Respiratory questionnaire
* Regional and widespread pain.
* Quality of life questionnaire.
* Most recent laboratory tests will be recorded (assessed in the HIV-negative cohort): renal, liver, lipid and bone profiles, glucose, full blood count, sexual health screen, hepatitis C serology (within the previous year)
* Blood (serum, plasma, and PBMC) and urine samples: stored for subsequent projects of the potential pathogenic mechanisms underlying age-related diseases. This will included assessment of vitamin-D and PTH
* Blood (plasma) will be collected for pharmacokinetic analysis (including but not limited to antiretroviral drug exposure)

  5 MRI Sub-study
* A sub-study will be conducted at the Severance Hospital site for participants equal to and over the age of 50 both HIV +ve (n=20) and HIV -ve (n=20). Matching criteria would be age, sexual orientation, and socio-economic status (i.e. insurance coverage status).

The study will comprise of three study visits:

1. Screening
2. Visit 1 (Baseline visit)
3. Visit 2 (Follow up visit after 2 years) The study visits will include the following assessments Blood (serum, plasma, and PBMC), urine, CSF and stool samples stored for future analysis (genetic polymorphism associated with neurocognitive dysfunction, CSF concentrations of antiretrovirals, biomarkers such as CSF neurofilament light (NFL) chain concentration, microbiome of stool, etc) Neurocognitive testing Lumbar puncture examination Cerebral MRI scan Respiratory function and cardiac function assessments

6 Withdrawal of subjects from study

Subjects are allowed to decline further participation in the study at any time. This will not affect their future care.

7 Study timelines

Recruitment and baseline visits (visit 1) will take place from months 1-12, with annual visits from months 13-24 (visit 2) and 25-36 (visit 3)

ELIGIBILITY:
Inclusion Criteria:

1. Older HIV-positive cohort (n=500):

   * documented HIV infection
   * age >50 years at study entry
   * Korean ethnicity
   * likely route of HIV acquisition via sexual exposure by male to male exposure
   * able to comprehend study patient information leaflet.
   * Virologically suppressed subjects Subjects with primary HIV infection are eligible and investigators are encouraged to recruit such subjects. Our target population (those infected with HIV via sexual routes of men who have sex with men) has been chosen as this group represent the vast majority of older HIV-positive individuals attending for care in Korea; analyses of other groups (e.g. injection drug users, those infected through blood/blood products and transgender individuals), who may have very different needs and outcomes, would likely be under-powered.
2. Younger HIV-positive cohort (n=250):

   * documented HIV infection
   * age <50 at study entry*
   * Korean ethnicity
   * likely route of HIV acquisition via sexual exposure by male to male exposure
   * able to comprehend study patient information leaflet * this group will comprise of at least 70 subjects in each of the following age groups: 20-29, 30-39, 40-49 years. Recruitment will be monitored by the Study Monitoring Team
3. HIV-negative cohort (n=250):

   * documented negative HIV test at screening
   * age >50 years at study entry
   * Korean ethnicity
   * self reported sexual preferences of men who have sex with men

To enroll matched control, we will try to match age, sexual orientation, and participating clinic.

Exclusion Criteria:

* in the opinion of the investigator, those unable or unwilling to comply with the requirements of the study
* life expectancy less than 6 months

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects with primary HIV infection are eligible and investigators are encouraged to recruit such subjects. Our target population (those infected with HIV via sexual routes of men who have sex with men) has been chosen as this group represent the vast majority of older HIV-positive individuals attending for care in Korea; analyses of other groups (e.g. injection drug users, those infected through blood/blood products and transgender individuals), who may have very different needs and outcomes, would likely be under-powered.
Study Population: HIV infected population who visit the study hospitals (a tertiary care hospital and two secondary care hopitals) and HIV-noninfected population from community
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious medical conditions | 2 years
  • the incidence and presenting features of serious medical conditions such as coronary heart disease, stroke, renal disease, cancer and liver disease etc.
  thd diagnosis of serious medical conditions will be defined by the latest clinical diagnostic criteria for each serious medical conditions.
  For example,
  Coronary heart disease (CHD)/ Myocardial infarction (MI)
  Definitive MI:
  Evolving diagnostic ECG Or Diagnostic biomarkers
  Probable MI:
  Positive ECG findings plus cardiac symptoms or signs plus missing biomarkers, Or Positive ECG findings plus equivocal biomarkers.
  Possible MI:
  Equivocal biomarkers plus nonspecific ECG findings, Or Equivocal biomarkers plus cardiac symptoms or signs, Or Missing biomarkers plus positive ECG.

SECONDARY OUTCOMES:
Incidence of neurocognitive disease | 2 years
  Incidence of neurocognitive disease The incidence of neurocognitive disease will be determined by following assessment.
  1. A short patient questionnaire
  2. Staff administered neurocognitive testing
  3. Computerised cognitive testing
  Subjects will complete a detailed neuropsychological assessment measuring their functioning in cognitive domains known to be commonly affected by HIV. The Frascati criteria were used for diagnosing HAND, classified into asymptomatic neurocognitive impairment (ANI), minor neurocognitive disorder (MND) and HIV-associated dementia

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yong Choi, Principal Investigator — Division of Infectious Diseases, Department of Internal Medicine, Severance Hospital, Yonsei University Health System
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No